CLINICAL TRIAL: NCT03078699
Title: Prospective Ⅱ Study of Stereotactic Body Radiation Therapy for Thymoma and Thymic Carcinoma: Therapeutic Effect and Toxicity Assessment
Brief Title: Prospective Study of Stereotactic Body Radiation Therapy for Thymoma Inoma: Therapeutic Effect and Toxicity Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xueqin Yang, Clinical Professor, Third Military Medical University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PSSBRT
Record Dates: First submitted 2017-02-24; First posted 2017-03-13 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Thymoma; Thymic Tumor
Keywords: Thymoma; Thymic tumor; Stereotactic body radiotherapy
MeSH Terms: conditions — Thymoma; Thymus Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stereotactic body radiation therapy (Experimental)
  Interventions: Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — A total radiation dose of 35-50 Gy was delivered to the 50% isodose line covering at least 95% of the PTV (3.5-5Gy/fraction), and a total radiation dose of 49-70 Gy was delivered to the 70% isodose line covering at least 95% of GTV (4.9-7 Gy/fraction).
  Other Names: Gamma knife

SUMMARY:
For patients with unresectable or recurrent disease, radiation is routinely administered, often in combination with systemic chemotherapy. However, because of wide range of radiation, more complications of conventional radiotherapy limit its treatment dose. The local recurrence rates of conventional radiotherapy are dissatisfied.Stereotactic body radiation therapy(SBRT) well solved the problem above. On the one hand, by improving the single dose, it not only shortens the total radiation treatment, but also increases the total dose of equivalent biological effects.

DETAILED DESCRIPTION:
Thymoma is mainly divided into two types, invasive and noninvasive type, and more than 60% of patients belong to noninvasive thymoma. When feasible, complete surgical resection is the primary treatment. There are quite a number of thymoma patients that has lost its surgical indications when diagnosed. Even after complete resection, the recurrence rate can be about 20%. For patients with unresectable or recurrent disease, radiation is routinely administered, often in combination with systemic chemotherapy. However, because of wide range of radiation, more complications of conventional radiotherapy limit its treatment dose. The local recurrence rates of conventional radiotherapy are up 16% to 45%. Moreover, it's not suitable for patients with severe heart and lung disease. Stereotactic body radiation therapy(SBRT) well solved the problem above. On the one hand, by improving the single dose, it not only shortens the total radiation treatment, but also increases the total dose of equivalent biological effects; On the other hand, SBRT, with more precise conformal radiation therapy, significantly reduces the damage to the surrounding normal tissues. Theoretically, SBRT can improve the local control, as well greatly reduces incidence of the radiation pneumonia, pericarditis, tracheitis, esophagitis and so on. However, few studies focused on the treatment of thymoma by SBRT, except two case reports Here we performed a prospective study on the treatment of thymoma by SBRT. The purpose of this prospective study was a preliminary evaluation of feasibility, efficacy and toxicity ofγ-SBRT in the treatment of thymoma.

ELIGIBILITY:
* Inclusion Criteria: Histologic or cytologic diagnosis of thymoma, Stage II-IV.

  * Males or females between 18 Years to 75 Years.
  * No prior SBRT, if the surgery or chemotherapy has been administered, the interval is at least above four weeks.
  * Performance status of 0, 1 on the ECOG criteria. Expected survival is above three months.
  * At least one unidimensional measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST. 2000).
  * Patients can have the brain / meningeal metastasis history, but the metastasis must be treated by operation or radiotherapy), and clinically stable for at least 2 months.
  * Adequate hematologic (neutrophil count >= 1,500/uL, platelets >= 100,000/uL), hepatic (transaminase =< upper normal limit(UNL)x2.5, bilirubin level =< UNLx1.5), and renal (creatinine =< UNL) function.
  * Patient compliance that allow adequate follow-up. Informed consent from patient or patient's relative.
  * If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 2 months after trial. If male, use of an approved contraceptive method during the study and 2 months afterwards. Females with childbearing potential must have a urine negative HCG test within 7 days prior to the study enrollment.
  * No concomitant prescriptions including cyclosporin A, valproic acid, phenobarbital, phenytoin, ketoconazole.
* Exclusion Criteria:

  * No pathological or cytological evidence of cancer.
  * Inability to comply with protocol or study procedures.
  * Medically uncontrolled serious heart, lung, neurological, psychological, metabolic disease Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
  * Pregnant or breast-feeding.
  * Enrollment in other study within 30 days.
  * Brain metastasis with symptoms.
  * Hypokalemic and intestinal obstruction history.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
PFS (progression-free time) | measured from the start of SBRT until any area in recurrence or distant metastasis, assessed up to 1 years
Tumor response rate | the ratio between the number of responders and number of patients assessable for tumor response，assessed up to 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baschnagel AM, Mangona VS, Robertson JM, Welsh RJ, Kestin LL, Grills IS. Lung metastases treated with image-guided stereotactic body radiation therapy. Clin Oncol (R Coll Radiol). 2013 Apr;25(4):236-41. doi: 10.1016/j.clon.2012.12.005. Epub 2013 Jan 24. PMID 23352916
- [Background] Lee CM, Lee JD, Hobson-Webb LD, Bedlack RS, Salama JK. Treatment of Thymoma-Associated Myasthenia Gravis With Stereotactic Body Radiotherapy: A Case Report. Ann Intern Med. 2016 Aug 16;165(4):300-1. doi: 10.7326/L15-0469. Epub 2016 Mar 15. No abstract available. PMID 26974367